CLINICAL TRIAL: NCT06505876
Title: Effect of Oral Feeding on Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Study
Brief Title: Effect of Oral Feeding on Patients With Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chao Phya Abhaibhubejhr Hospital (Other Government)
Responsible Party: Principal Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Oral feeing-COPD
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Tube Feeding+Basic treatment (Experimental): The patients were provided with 1) basic treatment including intracranial pressure reduction, anti-infection therapy, blood pressure and blood glucose control.
  For the observation group, the nasogastric tube was removed, and Intermittent oro-esophageal tube feeding was initiated for nutrition support within 4 hours after completing the admission assessment, following the standard Intermittent oro-esophageal tube feeding procedure.
  Interventions: Behavioral: Basic treatment; Device: Oral Tube Feeding
- Nasogastric Tube Feeding+Basic treatment (Active Comparator): The patients were provided with 1) basic treatment including intracranial pressure reduction, anti-infection therapy, blood pressure and blood glucose control.
  Patients in the control group were provided with nutrition support by the indwelling nasogastric tube. The entire feeding process strictly followed the standardized procedure for nasogastric feeding.
  Interventions: Behavioral: Basic treatment; Device: Nasogastric Tube Feeding

INTERVENTIONS:
Behavioral: Basic treatment — including anti-infection therapy, blood pressure and blood glucose control
Device: Oral Tube Feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Oral Tube Feeding+Basic treatment
Device: Nasogastric Tube Feeding — The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: Nasogastric Tube Feeding+Basic treatment

SUMMARY:
This is a prospective, randomized controlled clinical trail that involved patients with Chronic Obstructive Pulmonary Disease.The goal of this clinical trial is to compare the clinical effect of Oral Tubes vs Nasogastric Tubes in patients with Chronic Obstructive Pulmonary Disease. The main questions it aims to answer are:

Compared to Nasogastric Tube Feeding, can the Oral esophageal Tube Feeding better improve the nutritional status and pulmonary infection

DETAILED DESCRIPTION:
This is a prospective, randomized controlled clinical trail that involved patients with Chronic Obstructive Pulmonary Disease.The goal of this clinical trial is to compare the clinical effect of Oral Tubes vs Nasogastric Tubes in patients with Chronic Obstructive Pulmonary Disease. The main questions it aims to answer are:

Compared to Nasogastric Tube Feeding, can the Oral esophageal Tube Feeding better improve the nutritional status and pulmonary infection

Participants will be divided into two groups randomly, with different nutritional support respectively.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD confirmed by spirometry
* ≥18 years of age
* Sinus rhythm ≥50/min and < 120/min at inclusion
* Written informed consent

Exclusion Criteria:

* Known hypersensitivity to metoprolol or related derivatives
* Sinus bradycardia (resting heart rate < 50/min)
* Sick sinus syndrome unless treated with a pacemaker
* Atrial fibrillation/flutter
* Clinical signs or previous diagnosis of heart failure, angina pectoris, myocardial infarction, cerebrovascular disease, or critical peripheral ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Chronic Obstructive Pulmonary Disease Assessment Test | day 1 and day 15
  It is a simple questionnaire used to assess symptoms and quality of life in patients with Chronic Obstructive Pulmonary Disease (COPD). The scale consists of 8 items covering the most common symptoms and impacts on quality of life in COPD patients, such as cough, sputum production, and breathlessness. Each item is graded on a scale of 0 to 5, where patients select the score that best reflects their experience. The total score ranges from 0 to 40, with higher scores indicating more severe symptoms.